CLINICAL TRIAL: NCT05047718
Title: Factors Influencing the COVID-19 Vaccine Immune Response (Reactogenicity and Immunogenicity) According to Age and Presence or Not of a Past History of COVID-19
Brief Title: Factors Influencing the COVID-19 Vaccine Immune Response According to Age and Presence or Not of a Past History of COVID-19
Acronym: COVIMMUNAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Bioster, a.s. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21CH134; 2021-003547-24 (EudraCT Number)
Record Dates: First submitted 2021-09-14; First posted 2021-09-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Immunogenicity; reactogenicity; mRNA COVID-19 vaccine; COVID-19 natural immunity; age
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- convalescent participants PFIZER (Experimental): Participants with prior history of COVID-19 in ≥3 months, virologically confirmed and vaccinated by anti-covid19 Pfizer vaccine
  Interventions: Biological: COVID-19 vaccine Pfizer (2 doses)
- Naive participants PFIZER (Experimental): Participant without past history of COVID-19 and vaccinated by anti-covid19 Pfizer vaccine
  Interventions: Biological: COVID-19 vaccine Pfizer (3 doses)
- convalescent participants MODERNA (Experimental): Participants with prior history of COVID-19 in ≥3 months, virologically confirmed and vaccinated by anti-covid19 Moderna vaccine
  Interventions: Biological: COVID-19 mRNA Vaccine Moderna (2 doses)
- Naive participants MODERNA (Experimental): Participant without past history of COVID-19 and vaccinated by anti-covid19 Moderna vaccine
  Interventions: Biological: COVID-19 mRNA Vaccine Moderna (3 doses)
- Boost only (Experimental): Participant without past history of COVID-19 and vaccinated by anti-covid19 mRNA vaccine.
  Interventions: Biological: COVID-19 mRNA Vaccine Moderna (1 dose)

INTERVENTIONS:
Biological: COVID-19 vaccine Pfizer (3 doses) — A longitudinal analysis of the immune response post COVID-19 vaccine will be performed with a close immunomonitoring
  Arms: Naive participants PFIZER
Biological: COVID-19 vaccine Pfizer (2 doses) — A longitudinal analysis of the immune response post COVID-19 vaccine will be performed with a close immunomonitoring
  Arms: convalescent participants PFIZER
Biological: COVID-19 mRNA Vaccine Moderna (3 doses) — A longitudinal analysis of the immune response post COVID-19 vaccine will be performed with a close immunomonitoring
  Arms: Naive participants MODERNA
Biological: COVID-19 mRNA Vaccine Moderna (2 doses) — A longitudinal analysis of the immune response post COVID-19 vaccine will be performed with a close immunomonitoring
  Arms: convalescent participants MODERNA
Biological: COVID-19 mRNA Vaccine Moderna (1 dose) — A longitudinal analysis of the immune response post COVID-19 vaccine will be performed with a close immunomonitoring
  Arms: Boost only

SUMMARY:
Age is the main risk factor associated with the severity of COVID-19. From the beginning of the vaccination campaign, elderly subjects are part of the priority population. However, immunosenescence appears to play a role in the natural post-COVID-19 immunity of convalescent elderly subjects and also in the post-vaccination response. However, vaccination recommendations for both naïve (2 doses of vaccine) and convalescent subjects (1 dose of vaccine) do not differ according to age. To date, there is little data to suggest that the response to the vaccine in naïve or convalescent subjects may vary according to age in terms of qualitative and quantitative response and duration.

DETAILED DESCRIPTION:
In addition, the reactogenicity following the vaccine, remains important with COVID-19 vaccines, whether using an Messenger RiboNucleic Acid (mRNA) technique or an adenovirus vector technique. A better understanding of the parameters of early inflammatory response explaining this reactogenicity would allow to optimize the formulation of future vaccines. There are still several unknowns concerning the post-vaccination immune response (immunogenicity and reactogenicity) in older subjects,depending on their history of COVID-19 and the type of vaccine administered. A better understanding of this immune response is necessary in order to propose the best vaccine strategies and regimens in this high-risk COVID-19 population.

Thus, in partnership with Sanofi Pasteur and Bioaster, the Group On Mucosal Immunity And Pathogens (GIMAP) and Circulating Immune Complexes (CIC) vaccinology team proposes to conduct a study comparing the humoral, cellular, mucosal and reactogenic post-vaccination immune response in subjects with a history of COVID-19 >3 months ago (convalescent, 1 dose of vaccine) versus subjects with no history of COVID-19 (naive, 1 or 2 doses of vaccine depending on the type of vaccine used) according to age.

ELIGIBILITY:
Inclusion Criteria:

* For the group with a past history of COVID-19 (convalescents)= subject within ≥ 3 months after infection
* For the NO past history of COVID-19 (naives), subject with no known history of COVID-19
* Patient affiliated or entitled to a social security plan
* Patients who have received informed information about the study and who have co-signed a consent to participate in the study with the investigator

Exclusion Criteria:

* Immunocompromised or under immunosuppressive treatment
* Subject with a history of COVID hospitalized in intensive care
* Subject allergic to one of the components of the vaccines used in the study
* subject vaccinated for COVID-19
* Subject with persistent symptoms of COVID-19 (long COVID)
* Subjects with unstable chronic pathology
* Persons deprived of liberty, hospitalized without consent
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Anti-S neutralizing antibody titer | Days : 15, 90, 180 after each dose of vaccine
  The neutralizing antibody titer against protein S from the majority variants at the time of sampling and vaccine S will be evaluated in viral neutralization and pseudoneutralization

SECONDARY OUTCOMES:
Kinetic of Anti-S antibody titer | Days : 15, 90, 180 after each dose of vaccine
  The antibody titer against protein S will be evaluated by ELISA
Kinetic of Anti-N antibody titer | Days : 15, 90, 180 after each dose of vaccine
  The antibody titer against protein N will be evaluated by ELISA
Kinetic of Anti-SARS-CoV-2 immunoglobulin A (IgA) titers in saliva | Days : 15, 90, 180 after each dose of vaccine
Kinetic of SARS-CoV-2 quantiferon value | Days : 15, 90, 180 after each dose of vaccine
CD4 and CD8 lymphocyte polarization specific to the vaccine S protein | Days : 15 (group Naive and convalescent), 180 (group Boost only) after last dose of vaccine
  Evaluate by TruCulture (Myriad) methode
Anti-S neutralizing antibody titer | Days : 15, 90, 180 after each dose of vaccine
  The neutralizing antibody titer against protein S from the majority variants at the time of sampling and vaccine S will be evaluated in viral neutralization and pseudoneutralization
Kinetic of serum cytokine levels | At 24 and 72 hours after each dose of vaccine
Kinetic of C-reactive protein | At 24 and 72 hours after each dose of vaccine
Kinetic of vaccine-induced genes signatures | At 24 and 72 hours after each dose of vaccine
  Expression kinetics in foldchange (transcriptomics) of vaccine-induced gene signatures in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth BOTELHO-NEVERS, MD PhD, Principal Investigator — CHU de St Etienne
Locations (2):
- France (2):
  - HCL - Hôpital Croix Rousse, Lyon
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No